CLINICAL TRIAL: NCT02134860
Title: A Randomized Controlled Study on the Incretin Effect, Cognitive Function and Controlled Fasting During Bed Rest in Healthy Male Volunteers
Brief Title: Bed Rest, Alternate Daily Fasting and Incretin Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-6-2014-017
Record Dates: First submitted 2014-04-29; First posted 2014-05-09 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes; Critical Illness
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Critical Illness | interventions — Bed Rest; Glucose Tolerance Test; Neuropsychological Tests; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isocaloric diet (Active Comparator): 3 daily meals
  Interventions: Other: Bed rest; Other: OGTT; Other: IVGTT; Other: Cognitive testing; Other: Muscle and fat biopsies; Other: Dual-energy X-ray Absorptiometry (DXA) scan; Other: MRI
- Alternate daily fasting (Active Comparator): One meal (25% of caloric need) every second day and four meals (175% of caloric need) every second day
  Interventions: Other: Bed rest; Other: OGTT; Other: IVGTT; Other: Cognitive testing; Other: Muscle and fat biopsies; Other: Dual-energy X-ray Absorptiometry (DXA) scan; Other: MRI

INTERVENTIONS:
Other: Bed rest — 8 days of full bed rest
Other: OGTT — Oral glucose tolerance test with 75 g of glucose before and after bed rest
Other: IVGTT — Intravenous glucose tolerance test mimicking the glucose profile from the corresponding OGTT
Other: Cognitive testing — Daily testing of memory and concentration using standardized tests
Other: Muscle and fat biopsies — Biopsies will be obtained before and after bed rest
Other: Dual-energy X-ray Absorptiometry (DXA) scan — DXA scan to evaluate fat and muscle distribution before and after bed rest
Other: MRI — Functional MRI to evaluate cognitive function and abdominal MRI to evaluate visceral fat before and after bed rest

SUMMARY:
Bed rest produces insulin resistance in healthy volunteers. In this study the investigators aim to investigate the effect of 8 days bed rest on the incretin effect and how alternate daily fasting affects cognitive function and the insulin resistance produced by bed rest.

The subjects will be randomized to either 3 meals a day (isocaloric diet), alternate daily fasting or one meal/day every second day (25% of daily calorie need) and four meals/day every second (175% of daily calorie need).

The investigators hypothesize:

1. Bed rest reduces the incretin effect
2. Alternate daily fasting improves the cognitive function (memory and concentration) compared to isocaloric diet
3. Alternate daily fasting reduces insulin resistance produced by bed rest compared to isocaloric diet

DETAILED DESCRIPTION:
All subjects will undergo 8 days of bedrest. Outcome measures will be performed before, under and immediately after the bed rest period.

The individual study period will be 10 days in total.

ELIGIBILITY:
Inclusion Criteria:

* BMI<25kg/m2
* VO2 max normal for age

Exclusion Criteria:

* Tobacco smoking
* Alcohol ingestion > 14 units per week
* Diabetes in nearby relatives
* Resection of the small intestine
* History of gastric bypass surgery
* Risk of deep venous thrombosis
* Female

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incretin effect | 24 weeks
  Measured by Insulin levels during Oral glucose tolerance test (OGTT) and Intravenous glucose tolerance test (IVGTT)
Cognitive function | 18 months
  Evaluated by cognitive testing and functional Magnetic Resonance imaging (MRI)
Insulin resistance | 12 weeks
  Evaluated by insulin resistance indexes, HOMA-IR and Matsuda index

CONTACTS AND LOCATIONS:
Overall Officials: Nina Majlund Harder-Lauridsen, MD, Principal Investigator — Rigshospitalet, 7641; Signe Tellerup Nielsen, MD, Principal Investigator — Rigshospitalet, 7641; Rikke Krogh-Madsen, MD. PhD, Principal Investigator — Rigshospitalet, 7641; Bente Klarlund Pedersen, Professor, Study Director — Rigshospitalet, 7641
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717